CLINICAL TRIAL: NCT05750017
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate Safety and Tolerability of a Recombinant Herpes Zoster Vaccine (LZ901) in Subjects Aged 50 to 70 Years Inclusive
Brief Title: A Study to Evaluate Safety and Tolerability of a Recombinant Herpes Zoster Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Luzhu Biotechnology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LZ901-1
Record Dates: First submitted 2023-02-09; First posted 2023-03-01 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Herpes Zoster; Vaccine-Preventable Diseases
Keywords: Herpes Zoster; Vaccine
MeSH Terms: conditions — Herpes Zoster; Vaccine-Preventable Diseases | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort1: Low dose sentinel group (Experimental): Three subjects will be first enrolled into low dose sentinel group in open-label, prior to initiation of dosing in each dose level main group.
  Interventions: Biological: Low Dose Recombinant Herpes Zoster Vaccine (LZ901)
- Cohort2: High dose sentinel group (Experimental): After reviewing the safety through 7 days after the first dose of LZ901, if no safety signals occur, another 3 subjects will be enrolled into high dose sentinel group in open-label.
  Interventions: Biological: High Dose Recombinant Herpes Zoster Vaccine (LZ901)
- Cohort3: Low dose main group (Placebo Comparator): If also no safety signals occur through 7 days after the first dose of LZ901 in high dose sentinel group, 30 subjects will be randomized in a 2:1 ratio to receive two doses of LZ901 or placebo in a double-blind fashion in low dose main group.
  Interventions: Biological: Low Dose Recombinant Herpes Zoster Vaccine (LZ901); Drug: Placebo
- Cohort4: High dose main group (Placebo Comparator): Subjects will be enrolled in high dose main group also after the safety review through 7 days after the first dose of LZ901 or placebo in low dose main group.
  Interventions: Biological: High Dose Recombinant Herpes Zoster Vaccine (LZ901); Drug: Placebo

INTERVENTIONS:
Biological: Low Dose Recombinant Herpes Zoster Vaccine (LZ901) — 0.5 mL per dose, containing a total of 50 µg recombinant herpes zoster virus glycoprotein E, adjuvanted with alumina adjuvant.
  Arms: Cohort1: Low dose sentinel group; Cohort3: Low dose main group
Biological: High Dose Recombinant Herpes Zoster Vaccine (LZ901) — 0.5 mL per dose, containing a total of 100 µg recombinant herpes zoster virus glycoprotein E, adjuvanted with alumina adjuvant.
  Arms: Cohort2: High dose sentinel group; Cohort4: High dose main group
Drug: Placebo — 0.5 mL per dose, containing 4.5 mg sodium chloride.
  Other Names: Saline solution
  Arms: Cohort3: Low dose main group; Cohort4: High dose main group

SUMMARY:
This clinical trial is to study the safety and tolerability of a recombinant herpes zoster vaccine (LZ901) and sponsored by Beijing Luzhu Biotechnology Co., Ltd. It is a phase I, randomized, double-blind, placebo-controlled, dose escalation study in healthy people aged 50 to 70 years inclusive. The study is to protect adults against shingles (herpes zoster / varicella zoster virus(VZV)). There will be about 66 participators who will receive two-dose injection at the upper arm.

LZ901 vaccine is made up of a tetramer of VZV glycoprotein E (VZV gE-Fc) and adsorbed with aluminum hydroxide adjuvant. This adjuvant can raise the immune response to a lot of antigens. It is the most widely used and safe adjuvant in various types of vaccines worldwide.

In this study:

1. The participation is voluntary.
2. Before the study, participants will receive some tests for screening. If qualified, investigators will officially invite them to join this study.
3. The study vaccine is LZ901 with two different dose levels (50μg/0.5 mL, 100μg/0.5 mL). The placebo, which is saline solution, has no active drug. Participants will receive one of three as above mentioned.
4. Participants will be enrolled in one of four cohorts. If participants are enrolled in Cohorts 1 or 2, they will receive LZ901. If participants are enrolled in Cohorts 3 or 4, they will have a 2 out of 3 chance (66%) of receiving LZ901 and 1 out of 3 chance (33%) of receiving placebo.
5. In Cohort 3 and 4, the study staff and participants will not know which study treatment participants will be receiving. However, the study doctor can get this information in case of an emergency.
6. Participants will stay at the clinic for 30 minutes after each vaccination to observe if there are any uncomfortable.
7. This study will last about 8 months and will include about 8 study visits to the clinic. During this period, participants will receive a follow-up phone call and/or email by the study staff to follow the condition closely for safety, and record on diary/contact card.
8. Participants will receive some tests during the study, include safety tests such as physical examination, vital signs measurements, blood tests, urinalysis. Participants will be measured the levels of specific antibodies to see if the vaccine works well.

This study is for research purposes only. Participants may not receive any direct benefits from participating in this study but have a chance to be in a study that may help others in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females able to provide legal identity certificate, aged 50 to 70 years inclusive at the time of signing the ICF;
2. Able to understand the study procedures, voluntarily agree to participate in the study, and sign the ICF;
3. Subjects are healthy or have well controlled mild medical conditions as determined by the investigator；
4. Female subjects are not pregnant or lactating. Female subjects with childbearing potential* should take reliable contraceptive measures**, and have no pregnancy and fertility plan within 7 months;

   *Female subjects of childbearing potential are defined as sexually mature women: 1) have not undergone hysterectomy, bilateral salpingectomy, and bilateral oophorectomy; 2) have had natural menses at any time in the preceding 12 consecutive months (without an alternative medical cause). Post-menopausal should be confirmed with FSH and Estradiol levels.

   **Reliable, medically acceptable forms of contraception:
   * For 3 months prior to screening - hormonal contraceptive (e.g., oral, patch, injectable, depot or vaginal ring), or implantable device (implantable rod or intrauterine device), or
   * For at least 1 month prior to screening - a double barrier method (e.g., diaphragm, cervical cap, or condom in conjunction with spermicide or sponge), or
   * Subjects of reproductive age that are abstinent are acceptable provided they agree to a double barrier method should they become sexually active during the study.
   * and subjects agree to continue birth control for at least 7 months.
5. Able to attend all scheduled follow-up visits and able to comply with protocol requirements;
6. Oral temperature < 37.5℃/99.5℉.

Exclusion Criteria:

1. Subjects with a personal history or family history of convulsion, epilepsy, encephalopathy, and psychosis;
2. Subjects who received immunosuppressive therapy within 3 months before vaccination (e.g., long-term use of systemic glucocorticoids for ≥ 14 days, dose ≥ 2 mg/kg/day or ≥ 20 mg/day prednisone or equivalence);
3. Allergic to any component of the investigational vaccine, or have a history of a severe allergy to any vaccination;
4. Impaired immune function or diagnosed with congenital or acquired immunodeficiency disease, positive serology for Hepatitis B Surface Antigen, Hepatitis C Antibody and human immunodeficiency virus (HIV);
5. History of varicella or herpes zoster vaccination;
6. History of HZ;
7. Received an inactivated or recombinant vaccine within 14 days or any live vaccine within 28 days prior to vaccination;
8. Subjects who have acute diseases within 3 days before vaccination, or acute stage or exacerbation of chronic diseases within 1 month before vaccination;
9. Subjects with tattoos to the upper arm deltoid area or have infectious skin disease;
10. History of thrombocytopenia or other coagulation disorders, which may cause contraindications to intramuscular injection;
11. History of asplenia or functional asplenia, and asplenia or splenectomy due to any condition;
12. Subjects with ≥ Grade 2 laboratory abnormalities and Grade 1 laboratory abnormalities that the investigator consider clinically significant;
13. Participating in other clinical studies of investigational or un-registered products (drugs, vaccines or devices, etc.), or planning to participate in other clinical studies before the end of this clinical study;
14. Any conditions that in the opinion of the investigator may affect subject safety or assessments (disease factors such as extensive psoriasis, unexplained skin rash, eczema, chronic pain syndrome, or social factors such as plans to move elsewhere before the end of the study).
15. A positive screen for alcohol, drugs of abuse at screening period and Day 0 (before vaccination).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Solicited AEs | From Day 0 through Day 6 after each vaccination.
  A solicited AE is a pre-specified outcome that the subject is asked to record as present or not.
  The solicited AEs can be classified as vaccination site (local) AEs and Solicited systemic AEs based on the occurrence site.
Unsolicited AEs | From Days 0~29 after each vaccination.
  Unsolicited AEs include all AEs, except solicited AEs reported Days 0~6 after the study intervention.
AEs leading to withdrawal | From Day 0 until the outcome is clear after the following up, up to the end of study.
  The incidence of AEs leading subjects to withdrawal according to criteria for subject treatment discontinuation and withdrawal from study.
SAEs and MAAEs | From Day 0 through 6 months after the full course vaccination.
  The incidence of all serious adverse events (SAEs) and medically attended adverse events (MAAEs).
Abnormal laboratory tests results | On Day 3 (+ 1 day) after each study intervention.
  The incidence of abnormal laboratory tests results.

SECONDARY OUTCOMES:
The seropositivity rate of anti-gE antibody | On Day 30 after each study intervention.
  The percentage of seropositive subjects of anti-gE antibody.
The seropositivity rate of anti-VZV antibody | On Day 30 after each study intervention.
  The percentage of seropositive subjects of anti-VZV antibody.
Geometric mean concentration (GMC) of anti-gE | On Day 30 after each study intervention.
  Measured by ELISA.
Geometric mean titer (GMT) of anti-VZV | On Day 30 after each study intervention.
  Measured by fluorescent antibody to the membrane antigen (FAMA).
The seroconversion rate of anti-VZV antibody | On Day 30 after each study intervention.
  Seroconversion refers to at least a 4-fold increase in the anti-VZV antibody titer at the endpoint as compared to the prevaccination concentration (for subjects seropositive pre-vaccination) or a 4-fold increase at the endpoint as compared to the anti-VZV antibody titer cut-off value for seropositivity (for subjects seronegative pre-vaccination).
The seroconversion rate of anti-gE antibody | On Day 30 after each study intervention.
  Seroconversion refers to at least a 4-fold increase in the anti-gE Ab concentration at the endpoint as compared to the prevaccination concentration (for subjects seropositive pre-vaccination) or a 4-fold increase at the endpoint as compared to the anti-gE Ab cut-off value for seropositivity (for subjects seronegative pre-vaccination).
Change of anti-Fc antibody | From pre-immunization to Day 30 after each study intervention.
  Change of anti-Fc antibody on Day 30 after each study intervention compared with pre-immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No